CLINICAL TRIAL: NCT04621487
Title: A Randomized Controlled Trial: Quadruple vs Tailored Therapy in the Treatment of Helicobacter Pylori Infection
Brief Title: Quadruple vs Tailored Therapy in the Treatment of Helicobacter Pylori Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 004/08-19-03
Record Dates: First submitted 2020-10-21; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Amoxicillin; Metronidazole; Clarithromycin; Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- concomitant (Active Comparator): Concomitant therapy consists of 14 days pantoprazole 40 mg, amoxicillin 1000 mg, clarithromycin 500 mg, metronidazole 500 mg all twice daily.
  Interventions: Drug: Amoxicillin; Drug: Metronidazole; Drug: Clarithromycin; Drug: Pantoprazole 40mg
- tailored (Active Comparator): Tailored therapy consists of 14 days antibiotic therapy according to H. Pylori strains antibiotic sensitivity test together with pantoprazole 40 mg twice daily.
  Interventions: Drug: according to antibiogram

INTERVENTIONS:
Drug: Amoxicillin — 14 days 1 gr bid
  Arms: concomitant
Drug: Metronidazole — 14 days 500 mg bid
  Arms: concomitant
Drug: Clarithromycin — 14 days 500 mg bid
  Arms: concomitant
Drug: Pantoprazole 40mg — 40 mg bid 14 days
  Other Names: Pantoprazole
  Arms: concomitant
Drug: according to antibiogram — according to antibiogram
  Arms: tailored

SUMMARY:
Non-bismuth quadruple therapies have been proposed as potential strategies in improving the efficacy of first-line treatments. The non-bismuth quadruple therapy in its concomitant variant consists of proton pump inhibitor, amoxicillin, nitroimidazole and clarithromycin given concurrently twice daily. As a result of concurrent administration this therapy has given better results according to some studies in comparison to sequential variants. However, this therapy, as well suffers from the aforementioned increase in antibiotic resistance. Therefore, the aim of this study was to compare concomitant non-bismuth quadruple therapy with a tailored therapy based on antibiotic strain susceptibility testing.

DETAILED DESCRIPTION:
More than half of world population are H.pylori carriers. The infection is mostly acquired in childhood and persists lifelong. A notable risk factor is a lower social and economic status during childhood reflecting mostly poor hygienic standard or small and dense living area. Newly acquired infections in adulthood are a rarity. The reservoir of H. Pylori is the human stomach. H. pylori is considered to be the main pathogen involved in causing benign peptic ulcer and functional dyspepsia as well as gastric cancer. The treatment of H. Pylori infection is currently complicated by an increase in antimicrobial resistance in different parts of the world. Corresponding increase in clarithromycin as well as quinolone and metronidazole resistance poses a major clinical problem and calls for a new approach to treatment. Under such circumstances there is an emerging trend towards personalized eradication therapy. Since H. Pylori infection is an infectious disease its optimal treatment should both theoretically and practically be based on the specific characteristics of the strain and if possible the host of the infection. The aim of such an approach should be a better eradication efficacy.

Non-bismuth quadruple therapies have been proposed as potential strategies in improving the efficacy of first-line treatments. The non-bismuth quadruple therapy in its concomitant variant consists of proton pump inhibitor, amoxicillin, nitroimidazole and clarithromycin given concurrently twice daily. As a result of concurrent administration this therapy has given better results according to some studies in comparison to sequential variants. However, this therapy, as well suffers from the aforementioned increase in antibiotic resistance. Therefore, the aim of this study was to compare concomitant non-bismuth quadruple therapy with a tailored therapy based on antibiotic strain susceptibility testing assuming that eradication rate with tailored therapy will be above 90%.

ELIGIBILITY:
Inclusion Criteria:

* helicobacter pylori infection

Exclusion Criteria:

* previous unsuccessful eradication treatment, stomach or other malignancy, taking of proton pump inhibitors, H2-antagonists, bismuth or antibiotics (amoxicillin, metronidazole, clarithromycin) in the previous month, significant comorbidities (renal insufficiency, psychiatric disease), denial to participate in the study, history of allergy to proton pump inhibitors or antibiotics, pregnancy and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
eradication | 1 month after finishing therapy
  H.pylori status will be tested 1 month after therapy with a stool antigen test: positive or negative

SECONDARY OUTCOMES:
compliance | 1 month after finishing therapy
  compliance will be measured by counting pills that were taken during therapy, more than or equal to 80% will be considered as good compliance
adverse event | 1 month after finishing therapy
  patients will be asked to report any adverse events that occurred during treatment, they will be divided in groups, according to the degree of limitation of daily activities: no adverse events, mild (no limitations of activities), moderate (partially limited activities), severe (completely limited)

CONTACTS AND LOCATIONS:
Overall Officials: Nikola Perkovic, MD, Principal Investigator — University Hospital of Split
Locations (1):
- University hospital Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: No